CLINICAL TRIAL: NCT04237142
Title: Preterm Premature Rupture of Fetal Membranes: Cervical Ultrasound and Biological Markers to Diagnose Prematurity.
Brief Title: Preterm Premature Rupture of Fetal Membranes: Cervical Ultrasound and Biological Markers to Diagnose Prematurity (RECHOBIOL)
Acronym: RECHOBIOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Biosynex Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2019 GALLOT; 2019-A02306-51 (Other: ANSM)
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Premature Rupture of Membrane
Keywords: Preterm premature rupture of membranes; Biomarkers; Latency period; Predictive Value of Tests
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes | interventions — Blood Specimen Collection

STUDY DESIGN:
Masking Description: Results of the biological tests are masked for the clinician and the patient and therefore do not modify the current management. Results will be given after delivery in order to not influence the current medical care of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients who had consented to participate (Experimental): Eligible patients who had consented to participate to the study, namely parturient admitted to the Clermont-Ferrand Hospital maternity for preterm premature rupture of membranes between 24+0 and 36+4 gestation week with cervical dilation < 4cm and without known uterine malformation, fetal malformation, placenta previa or abundant metrorrhagia. Patients underwent vaginal swabbing and blood sample collection at the admission.
  Interventions: Diagnostic Test: Vaginal secretions collection; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Vaginal secretions collection — Vaginal secretions are collected under speculum with a swab (10 seconds of impregnation of the swab). The swab is immersed in a tube containing an extraction buffer for 10 seconds. The tube is mixed and sent to the laboratory for subsequent analysis of biomarkers (IGFBP1 T/N, PIBF, PP14) and storage.
Diagnostic Test: Blood sample — 2 tubes of blood sample were collected and sent to the laboratory for serum storage and biomarkeurs assay (PIBF and MIF)

SUMMARY:
Our main hypothesis is to consider that the detection of biomarkers on admission combined with the length of the cervix would improve the prediction of the latency period in case of preterm premature rupture of membranes (pPROM). The primary purpose of the protocol is to assess the performance of these tests to predict a latency period <48 hours in case of pPROM.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (pPROM) is defined as a spontaneous rupture before the start of labor ("premature" rupture) and before 37 weeks of gestation ("preterm"). pPROM concern 2-3% of pregnancies. It is the main cause of prematurity since it is responsible for 24 to 42% of preterm deliveries. The time between PROM and childbirth is named the latency period. Its total duration can vary from a few hours to several weeks. Childbirth occurs within 48 hours of rupture for 18 to 93% of cases, within 7 days for 56 to 96% and within 28 days for 78 to 100%. The earlier PROM occurs during pregnancy, the longer the latency period is. The factors associated with a shorter latency period are: cervical changes during admission for pPROM, a shortened cervix on ultrasound or a threat of premature delivery prior to PROM, the existence of uterine contractions, oligoamnios, and the occurrence of a materno-fetal complication of pPROM.

In a pPROM situation, a prolonged latency period improves the neonatal prognosis by increasing the gestational age of birth, gives the possibility of administering the corticosteroid treatment of fetal pulmonary maturation and also allows an in utero transfer in an adapted maternity.

Several studies have shown a correlation between the length of the cervix during rupture and the latency period in the context of pPROM.

To date, there are no effective biomarkers used in current practice to predict this latency period.

We want to assess the diagnostic performance of different vaginal (PIBF / PP14 / IGFBP1 native and total) and serum (PIBF / MIF) markers as well as the ultrasound length of the cervix to predict the duration of this latency period in order to better anticipate the risk of prematurity.

ELIGIBILITY:
Inclusion Criteria:

* Parturient admitted to the Clermont-Ferrand Hospital maternity for preterm premature rupture of membranes between 24+0 and 36+4 gestation week.
* Capacity to give informed consent.
* Coverage by a French social security scheme.

Exclusion Criteria:

* Refusal to participate
* pPROM formally occurred more than 24 hours ago (free flow or positive breakage test)
* Cervical dilatation ≥ 4 cm
* Multiple Pregnancy
* Known uterine malformation
* Fetal Malformation
* Placenta previa
* Abundant metrorrhagia
* Patient under guardianship or curatorship

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
total IGFBP1 in vaginal secretion at admission | Day 0
  Results of the tests detecting total IGFBP1 (positive/ negative)
native IGFBP1 in vaginal secretion at admission | Day 0
  Results of the tests detecting native IGFBP1 (positive/ negative)
PP14 in vaginal secretion at admission | Day 0
  PP14 values in vaginal secretion at admission dosed using the ELISA technique
PIBF in vaginal secretion at admission | Day 0
  PIBF values in vaginal secretion at admission dosed using the ELISA technique
PIBF in maternal serum at admission | Day 0
  PIBF values in maternal serum at admission dosed using the ELISA technique
MIF in maternal serum at admission | Day 0
  MIF values in maternal serum at admission dosed using the ELISA technique
Ultrasound length of cervix measured at the admission | Day 0
  Length of cervix was maesured by ultrasound at the admission (millmeters)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Gallot, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France